CLINICAL TRIAL: NCT04578548
Title: An Exploratory, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of Orally Administered GLPG2737 for 52 Weeks, Followed by an Open-label Extension Period of 52 Weeks in Participants With Autosomal Dominant Polycystic Kidney Disease
Brief Title: A Study to Evaluate the Effects of GLPG2737 in Participants With Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was early terminated due to lack of efficacy.
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLPG2737-CL-203; 2019-003521-21 (EudraCT Number)
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-03

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- GLPG2737 During DB + During OLE (Experimental): Participants received 150 milligrams (mg) GLPG2737 capsules orally once daily for 52 weeks in the double-blind (DB) treatment period. Eligible participants were rolled over to an open-label extension (OLE) period to receive 150 mg GLPG2737 orally once daily for 52 weeks.
  Interventions: Drug: GLPG2737
- Placebo During DB + GLPG2737 During OLE (Placebo Comparator): Participants received placebo matched to GLPG2737 capsules orally once daily for 52 weeks in the DB treatment period. Eligible participants were rolled over to an OLE period to receive 150 mg GLPG2737 orally once daily for 52 weeks.
  Interventions: Drug: GLPG2737; Drug: Placebo

INTERVENTIONS:
Drug: GLPG2737 — Capsules administered orally
Drug: Placebo — Matching placebo capsules administered orally
  Arms: Placebo During DB + GLPG2737 During OLE

SUMMARY:
This is an exploratory, randomized, double-blind, placebo-controlled, parallel group, multicenter, proof of concept study (Phase 2a), evaluating orally administered GLPG2737 for a double-blind (DB) treatment period of 52 weeks and 4 weeks of follow up as well as an open-label extension (OLE) treatment period of 52 weeks and 4 weeks of follow-up, in participants with rapidly progressing ADPKD.

ELIGIBILITY:
Key Inclusion Criteria for the double-blind period of the study:

* Documented diagnosis of typical ADPKD, using the Ravine criteria (Ravine, et al., 1994).
* Rapidly progressive disease, defined as presence of all of the following:

  * Total Kidney Volume (TKV) >750 mL, as determined on imaging not older than 5 years before screening. If historical imaging is not available or older than 5 years, imaging can be performed during the screening period according to local clinical practice (that is, echography, magnetic resonance imaging [MRI])
  * Mayo ADPKD Classification Classes 1C to 1E.
* eGFR at screening between 30 to 90 milliliters per minute per 1.73 square meter (mL/min/1.73 m^2) for participants aged 18 to 40 years (inclusive), and between 30 to 60 mL/min/1.73 m^2 for participants aged 40 to 50 years.
* Blood pressure ≤ 150/90 millimeters of mercury (mmHg). In case a participant is treated for hypertension, she/he should be on a stable treatment regimen of antihypertensive therapy for at least 8 weeks prior to the screening visit, and during the screening period.

Key Inclusion Criteria for the OLE period of the study:

* Male and female participants who completed the 52-week double-blind treatment period on investigational product (IP).
* Participant, according to the investigator's judgment, may benefit from long-term treatment with GLPG2737.

Key Exclusion Criteria for the double-blind period of the study:

* Congenital absence of 1 kidney, or participant had a previous nephrectomy or has a transplanted kidney or a transplantation is planned in the foreseeable future.
* Administration of polycystic kidney disease-modifying agents (for example, tolvaptan, somatostatin analogues) or interventions (such as cyst aspiration or cyst fenestration) within 12 weeks prior to the screening visit and during the screening period. In case tolvaptan is not being administered, this should be because of e.g. non-availability, intolerance, or physician's clinical judgment.
* Any condition or circumstances that, in the opinion of the investigator, may make a participant unlikely or unable to complete the study or comply with study procedures and requirements (for example, unable to undergo magnetic resonance imaging (MRI) due to participant's weight exceeds the weight capacity of the MRI, ferromagnetic metal prostheses, aneurysm clips, severe claustrophobia, etc.).

Key exclusion criteria for the OLE period of the study:

* Clinically significant abnormalities detected on 12-lead electrocardiogram (ECG) of either rhythm or conduction, QTcF >450 ms, or long QT syndrome.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (20):
- Belgium (2):
  - Cliniques Universitaires St. Luc (UCL), Brussels
  - UZ Leuven, Leuven
- Czechia (3):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Vseobecna fakultni nemocnice v Praze, Prague
- Uniklinikum Dresden, Dresden, Germany
- Italy (4):
  - IRCSS Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Uni Campania L. Vanvitelli, Napoli
  - Fondazione Salvatore Maugeri IRCCS, Pavia
- Netherlands (3):
  - Amsterdam UMC, Amsterdam
  - UMCG, Groningen
  - Radboud UMC, Nijmegen
- Poland (3):
  - Specjalistyczne Centrum Medyczne SCM Spółka z o.o., Krakow
  - Szpital Kliniczny UM w Lodzi, Lodz
  - DaVita Sp. z o.o. Stacja Dializ, Warsaw
- Spain (4):
  - Fundacion Puigvert, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Nefrologia Clinica C.P., Madrid
  - Hospital Universitario Dr. Peset, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ron T. Gansevoort et al., 2022. The MANGROVE Phase 2 Trial: Study Design and Baseline Characteristics of Patients With Autosomal Dominant Polycystic Kidney Disease (ADPKD). Abstract (385) presented at the Annual Congress of the American Society of Nephrology, 3-Nov-2022 to 6-Nov-2022.
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with autosomal dominant polycystic kidney disease (ADPKD) were enrolled. The study was conducted at 20 sites in 7 countries i.e. Belgium, Czech Republic, Germany, Italy, Netherlands, Poland, and Spain. Out of these 20 activated sites, 3 sites did not enroll any participants. 89 participants were screened, out of which 66 were randomized.
Pre-assignment Details: Participants who met protocol eligibility criteria were assigned to GLPG2737 or placebo in the double-blind (DB) treatment period and open-label extension (OLE) period. The study was prematurely terminated on 02 March 2023, due to the lack of efficacy of GLPG2737, making the expected benefit-risk balance negative.
Groups:
- GLPG2737 During DB + During OLE: Participants received 150 milligrams (mg) GLPG2737 capsules orally once daily for 52 weeks in the DB treatment period. Eligible participants were rolled over to an OLE period to receive 150 mg GLPG2737 orally once daily for 52 weeks.
Period: Double-blind Treatment Period (52 Weeks)
Arm/Group | GLPG2737 During DB + During OLE | Placebo During DB + GLPG2737 During OLE
Started | 44 | 22
Completed | 41 | 20
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Non Compliance with study drug | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Open-Label Treatment Period (52 Weeks)
Arm/Group | GLPG2737 During DB + During OLE | Placebo During DB + GLPG2737 During OLE
Started | 39 (Not all participants who completed the DB treatment period entered the OLE treatment period.) | 20
Completed | 3 | 4
Not Completed | 36 | 16
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Study terminated by sponsor | 34 | 15

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS): All randomized participants who received at least one dose of study drug.
Groups:
- GLPG2737 During DB: Participants received 150 mg GLPG2737 capsules orally once daily for 52 weeks in the DB treatment period.
- Placebo During DB: Participants received placebo matched to GLPG2737 capsules orally once daily for 52 weeks in the DB treatment period.
- Total: Total of all reporting groups
Arm/Group | GLPG2737 During DB | Placebo During DB | Total
Number analyzed (Participants) | 44 | 22 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (6.3) | 39.6 (6.2) | 40.3 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 8 | 32
  Male | 20 | 14 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 2 | 11
  Not Hispanic or Latino | 35 | 20 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 44 | 22 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height-Adjusted Total Kidney Volume(htTKV) [Mean (Standard Deviation); unit: mL/m] — htTKV is used in participants with ADPKD disease to predict the onset of renal insufficiency. htTKV was calculated using TKV (in milliliter [mL]) obtained from magnetic resonance imaging (MRI) divided by height (in meter [m]). MRI Baseline: For MRI assessments, all non-missing values before the first study drug administration in the study +14 days (included) was considered as the primary baseline definition. Population: SAS. Participants with MRI baseline were analyzed.
  mL/m
    number analyzed (Participants) | 41 | 20 | 61
    (all) | 1069.18 (438.06) | 1439.23 (737.67) | 1190.51 (575.26)
Estimated Glomerular filtration rate (GFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — eGFR is a test that measures level of kidney function and determines your stage of kidney disease. eGFR was based on chronic kidney disease-Epidemiology (CKD-EPI) formula (2009) calculated from serum creatinine concentrations. eGFR was measured as milliliters per minute per 1.73 square meter (mL/min/1.73 m^2).
  mL/min/1.73 m^2 | 55.5 (16.3) | 51.6 (15.6) | 54.2 (16.1)

OUTCOME MEASURES:

1. Primary Outcome: DB Period: Mean Percent Change From MRI Baseline in htTKV
Description: htTKV is used in participants with ADPKD disease to predict the onset of renal insufficiency. htTKV was calculated using TKV (in mL) obtained from MRI divided by height (in m). MRI Baseline: For MRI assessments, all non-missing values before the first study drug administration in the study +14 days (included) was considered as the primary baseline definition. Results were derived by mean of the individual slopes (i.e. using all MRI performed between baseline and Week 52).
Time Frame: MRI Baseline up to Week 52
Population: Full Analysis Set (FAS): All randomized participants who received at least one dose of study drug.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | GLPG2737 During DB | Placebo During DB
Number analyzed (Participants) | 44 | 22
percent change | 8.18 [6.04 to 10.36] | 9.17 [6.05 to 12.38]
Statistical Analysis 1: Comparison: GLPG2737 During DB vs Placebo During DB; Based on a random coefficient regression model (linear slope model) on htTKV log-transformed values with time (in weeks) as a continuous variable, treatment, time-by-treatment interaction and a random intercept and slope. The treatment effect was determined by using estimated slopes for each treatment group on the basis of the time-by-treatment interaction term from the mixed model; Test type: Superiority; p = 0.606, Random coefficient regression model; Geometric Mean Difference = -0.91, 95% CI 2-sided [-4.34 to 2.64]

2. Primary Outcome: DB Period: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE is any untoward medical occurrence in a participant administered a study drug, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of the study drug, whether or not considered related to it. A serious adverse event (SAE) is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results a congenital anomaly/birth defect or other medically important event. A TEAE was defined as an AE observed after starting administration of the study drug until 30 days after last DB dose or 1 day before OLE dose, whichever occurred first.
Time Frame: From first dose to Week 56
Population: SAS
Measure: Number; unit: participants
Arm/Group | GLPG2737 During DB | Placebo During DB
Number analyzed (Participants) | 44 | 22
participants
  TEAEs | 44 | 22
  Serious TEAEs | 1 | 3

3. Secondary Outcome: DB Period: Mean Change From Baseline in eGFR
Description: The eGFR is a test that measures level of kidney function and determines the stage of kidney disease. eGFR was based on CKD-EPI formula (2009) calculated from serum creatinine concentrations. Results were derived by mean of the individual slopes (i.e. using data between baseline and Week 52).
Time Frame: Baseline up to Week 52
Population: FAS
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73 m^2
Arm/Group | GLPG2737 During DB | Placebo During DB
Number analyzed (Participants) | 44 | 22
mL/min/1.73 m^2 | -5.44 [-7.34 to -3.54] | -3.13 [-5.87 to -0.39]
Statistical Analysis 1: Comparison: GLPG2737 During DB vs Placebo During DB; Least-squares mean difference (95% CI) from a random coefficient regression model (linear slope model) on eGFR values with time (in weeks) as a continuous variable, the time-by-treatment interaction and a random intercept and slope. The treatment effect was determined by using estimated slopes for each treatment group on the basis of the time-by-treatment interaction term from the mixed model; Test type: Superiority; p = 0.171, Random coefficient regression model; Least-squares mean difference = -2.31, 95% CI 2-sided [-5.64 to 1.02]

4. Secondary Outcome: DB Period: Area Under the Plasma Concentration-Time Curve During a Dosing Interval (AUCtau) of GLPG2737 and Its Metabolite
Description: AUC0-tau described the area under the curve limited to the end of a dosing interval. The metabolite of GLPG2737 is M4.
Time Frame: Predose (within 30 minutes prior to dosing), 1, 1.5, 2, 3, 4, 5, 6, 7 hours post dose through Week 52
Population: Pharmacokinetic Analysis Set (PKAS): All randomized participants who received at least one dose of study drug for which plasma concentration data was available to facilitate development of the Population PK model and for whom the time of the dose on the days of PK sampling was known.
Measure: Geometric Mean (95% Confidence Interval); unit: nanogram* hour per milliliter (ng*h/mL)
Arm/Group | GLPG2737 During DB
Number analyzed (Participants) | 44
nanogram* hour per milliliter (ng*h/mL)
  GLPG2737 | 18500 [17500 to 19500]
  Metabolite M4 | 18700 [17400 to 20200]

5. Secondary Outcome: DB Period: Maximum Observed Plasma Concentration (Cmax) of GLPG2737 and Its Metabolite
Description: Cmax is the maximum observed plasma concentration of the drug. The metabolite of GLPG2737 is M4.
Time Frame: Predose (within 30 minutes prior to dosing), 1, 1.5, 2, 3, 4, 5, 6, 7 hours post dose through Week 52
Population: PKAS
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | GLPG2737 During DB
Number analyzed (Participants) | 44
ng/mL
  GLPG2737 | 1160 [1110 to 1220]
  Metabolite M4 | 873 [813 to 939]

ADVERSE EVENTS:
Time Frame: DB Period: From first dose to Week 56 OLE Period: From first dose to Week 56
Description: DB Period: SAS.
  OLE Period: All OLE enrolled participants who received one dose of study drug during the OLE period.
Groups:
- GLPG2737 During DB + During OLE: Participants received 150 mg GLPG2737 capsules orally once daily for 52 weeks in the DB treatment period. Eligible participants were rolled over to an OLE period to receive 150 mg GLPG2737 capsules orally once daily for 52 weeks.
- Placebo During DB + GLPG2737 During OLE: Eligible participants from Placebo DB were rolled over to an OLE period to receive 150 mg GLPG2737 capsules orally once daily for 52 weeks.
Arm/Group | GLPG2737 During DB + During OLE | Placebo During DB | Placebo During DB + GLPG2737 During OLE
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 3/44 | 3/22 | 2/20
Other Adverse Events (participants affected / at risk) | 44/44 | 22/22 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLPG2737 During DB + During OLE (N=44) | Placebo During DB (N=22) | Placebo During DB + GLPG2737 During OLE (N=20)
Hepatic cyst infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Renal cyst infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cyst rupture (General disorders) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLPG2737 During DB + During OLE (N=44) | Placebo During DB (N=22) | Placebo During DB + GLPG2737 During OLE (N=20)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aortic bruit (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Defect conduction intraventricular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 2 (3) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 2 (3) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (5) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 11 (44) | 8 (18) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Mediastinal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (7) | 2 (6) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (5) | 3 (3) | 0
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 2 (3) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 11 (21) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 1 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (7) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Renal cyst ruptured (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (4) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 4 (8) | 2 (2) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Albuminuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 4 (11) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal cyst haemorrhage (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 4 (4) | 2 (2) | 2 (2)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Renal pain (Renal and urinary disorders) | 8 (15) | 6 (19) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Skin depigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 4 (9) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (6) | 2 (3) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (5) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Acrodermatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperparathyroidism secondary (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Bacterial vulvovaginitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 21 (25) | 5 (5) | 1 (1)
Cystitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gardnerella infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastric infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatic cyst infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 8 (10) | 2 (3) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 10 (16) | 5 (7) | 2 (2)
Norovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Phlebitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Renal cyst infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (8) | 3 (3) | 5 (6)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Chillblains (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 2 (4) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post vaccination syndrome (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Traumatic renal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 4 (9) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 13 (16) | 4 (4) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 3 (3) | 3 (3) | 0 (0)
Haematuria traumatic (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema mucosal (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (4) | 1 (2) | 0 (0)
Peripheral swelling (General disorders) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 6 (10) | 2 (3) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 1 (1)
Rubber sensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (3) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Drug intolerance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (6) | 3 (4) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The early termination was decided due to the lack of efficacy of GLPG2737, making the expected benefit-risk balance negative.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT04578548/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT04578548/SAP_001.pdf